CLINICAL TRIAL: NCT05851547
Title: A Phase II Study of the Use of MRI-defined Focal Boosts With Stereotactic Body Radiotherapy for Localized Prostate Cancer
Brief Title: Dose Escalation For INtraprostatic LEsions
Acronym: DEFINE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Knight Therapeutics (USA) Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220698-01H
Record Dates: First submitted 2023-03-21; First posted 2023-05-09 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Prostatic Neoplasms
Keywords: Localized Prostate Cancer; Intermediate Risk; High Risk; Stereotactic Body Radiotherapy; External Beam Radiotherapy; Hypofractionation; Focal Boost; Microboost; Androgen Deprivation Therapy; Multiparametric magnetic resonance imaging
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate; Androgen Antagonists

STUDY DESIGN:
Intervention Model Description: Prostate radiotherapy of 27 Gy in 3 fractions to uninvolved regions, up to 39 Gy in 3 fractions to mpMRI-defined intraprostatic lesions, with concurrent/adjuvant androgen deprivation therapy (6 months intermediate risk, 24 months for high risk)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostate SBRT with Focal Boost and Androgen Deprivation Therapy (Experimental): Stereotactic body radiotherapy to 27 Gy in 3 fractions to uninvolved regions of the prostate glad and up to 39 Gy in 3 fractions to mpMRI-defined intraprostatic lesions, with concurrent/adjuvant androgen deprivation therapy (6 months for intermediate risk, 24 months for high risk)
  Interventions: Radiation: Prostate SBRT with Focal Boost; Drug: Triptorelin Injection

INTERVENTIONS:
Radiation: Prostate SBRT with Focal Boost — Prostate stereotactic body radiotherapy delivered to 27 Gy in 3 fractions on alternating days to uninvolved regions with up to 39 Gy in 3 fractions delivered to mpMRI-defined intraprostatic lesions
  Other Names: Ultrahypofractionated prostate radiotherapy with integrated microboost
Drug: Triptorelin Injection — Six months of androgen deprivation therapy for intermediate-risk localized prostate cancer and 24 months for high-risk localized prostate cancer
  Other Names: Androgen Deprivation Therapy

SUMMARY:
External beam radiotherapy combined with androgen deprivation therapy is a standard treatment option for localized prostate cancer. The current standard involves delivering radiotherapy uniformly throughout the prostate gland in daily fractions, five days per week, for approximately four weeks. In this study, radiotherapy will be delivered using an ultra-hypofractionated approach in three larger fractions on alternating days over one week Multiparametric magnetic resonance imaging will be used to guide focal dose escalation to parts of the gland harboring tumor, which could potentially reduce the risk of cancer recurrence compared to standard dose of radiotherapy. The aim of this study is to confirm that this approach can be delivered safely, that is, with rates of urinary and bowel side effects at 1 year of follow-up that are not significantly greater than the current standard.

DETAILED DESCRIPTION:
External beam radiotherapy (RT) in combination with androgen deprivation therapy (ADT) is a standard definitive treatment for localized prostate cancer. It confers long-term oncologic outcomes equivalent to those of radical prostatectomy. The current standard approach for prostate RT consists of uniform irradiation of the entire gland. This technique employs computed tomography (CT) images for planning, in which disease is not readily apparent. Multiparametric magnetic resonance imaging (mpMRI) of the prostate allows for accurate visualization of clinically significant tumour foci within the prostate gland. It thereby permits selective escalation of dose to tumours within the gland - a so-called focal boost or "microboost" - with the aim of improving treatment efficacy.

The current standard approach to prostate RT involves delivery of treatment in daily fractions, five days per week, over four weeks. Prostate cancer appears to exhibit an uncommon fractionation sensitivity among solid tumours. A consequence of this is that hypofractionation - that is, delivery of RT with larger fraction sizes - may further improve the therapeutic ratio. A number of large-scale studies have shown promise for an ultra-hypofractionated approach (that is, larger than 5-Gy fractions) in the treatment of localized prostate cancer.

There is an unmet need for innovations in radiotherapy that further reduce the risk of relapse without increasing toxicity or compromising health-related quality of life and that reduce the treatment burden. Both focal intraprostatic boosts - informed by mpMRI findings - and ultra-hypofractionation represent promising approaches to achieve this objective. To date, the optimal regimen that combines these two innovations remains to be explored. In this trial, we will investigate in a single-arm prospective cohort the safety of an mpMRI-defined focal boost technique with a convenient and radiobiologically compelling ultra-hypofractionated radiotherapy regimen (consisting of three fractionas delivered over one week) for localized unfavourable intermediate and high-risk localized prostate cancer.

This is a single-arm prospective trial conducted in patients with unfavourable intermediate-risk or high-risk localized prostate cancer. Treatment consists of ultra-hypofractionated intensity-modulated, image-guided prostate radiotherapy delivered to 27 Gy in 3 fractions (1 fraction per day every other day, over a 5 day period) to uninvolved regions, with up to 39 Gy in 3 fractions delivered to mpMRI-defined intraprostatic lesions, assuming normal tissue dosimetric criteria can be safely met. Radiotherapy will be combined with concurrent/adjuvant androgen deprivation therapy (6 months duration in patients with intermediate-risk disease and 24 months for patients with high-risk disease). There will be follow-up assessments for toxicity, quality of life, and biochemical control. The primary endpoint will be prevalence of grade ≥ 2 genitourinary or gastrointestinal toxicity at 12 months.

Primary Objective The primary objective is to determine whether, in a population of men with unfavourable intermediate-risk or high-risk localized prostate cancer receiving a combination of three-fraction ultra-hypofractionated RT and adjuvant androgen deprivation therapy, an mpMRI-defined focal boost can be delivered with acceptable GU and GI toxicity at 1 year of follow-up.

Secondary Objectives

The secondary objectives are to evaluate, in a population of men with unfavourable intermediate-risk or high-risk localized prostate cancer, the effects of an mpMRI-defined focal boost on:

* Health-related quality of life
* Biochemical disease-free survival

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Unfavourable intermediate-risk or high-risk localized disease
* Unfavourable intermediate-risk prostate cancer is defined as intermediate-risk prostate cancer [that is, no high-risk features and one or more intermediate-risk factors: T2b-T2c, Gleason 3+4 (grade group 2) or Gleason 4+3 (grade group 3), or PSA 10-20 μg/L] and one or more of the following: 2 or 3 intermediate-risk factors; Gleason 4+3 (grade group 3); ≥ 50% biopsy cores positive
* High-risk localized prostate cancer is defined as at least one of the following: T3a-T3b; Gleason ≥ 8 (grade group 4 or grade group 5); PSA > 20 μg/L
* 3 Tesla prostate MRI done no more than 12 months prior to enrollment
* ECOG performance status 0-2
* Age ≥ 18 years
* Written informed consent
* The participant has planned androgen deprivation therapy that meets one of the following criteria:
* Patients with intermediate-risk localized prostate cancer who have planned androgen deprivation therapy consisting of up to 6 months of triptorelin with or without bicalutamide; OR patients with high-risk localized prostate cancer who have planned androgen deprivation therapy consisting of up to 24 months of triptorelin with or without bicalutamide.
* Completion of all appropriate investigations prior to enrollment

Exclusion Criteria:

* Evidence of pelvic nodal metastases or distant metastases (AJCC Stage T1-4 N1 M0-1 or T1-4 N0 M1 disease)
* Discordance between pre-enrollment prostate MRI and prostate biopsy findings, defined as biopsy cores with Gleason Gleason ≥ 4+3 (grade group ≥ 3) adenocarcinoma with no corresponding tumour focus seen on MRI
* Androgen deprivation therapy commenced more than 60 days prior to enrollment
* Intention to electively treat the pelvic lymph nodes with radiotherapy
* Other active malignancy within the previous three years (except adequately treated nonmelanomatous carcinoma of the skin or low-grade superficial bladder carcinoma)
* Prior pelvic radiotherapy
* Contraindication to pelvic radiotherapy
* Any history, past or present, of inflammatory bowel disease
* Unilateral or bilateral hip arthroplasty
* Trans-urethral resection of the prostate (TURP) performed within 6 months of anticipated start date of radiotherapy
* Patients must not concurrently participate in any other therapeutic prostate cancer trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Genitourinary and gastrointestinal toxicity | Up to 2 years
  Number of patients with grade 2 or greater genitourinary or gastrointestinal toxicity as measured by Common Terminology Criteria for Adverse Events (CTCAE ) version 5.0 and Radiation Therapy Oncology Group radiation toxicity scale

SECONDARY OUTCOMES:
Bowel and urinary quality of life | Up to 2 years
  Measured by Expanded Prostate Cancer Index Composite (EPIC)-26 bowel and urinary domains
Disease-free survival | 2 years
  Number of patients free of biochemical recurrence (defined according to the Phoenix definition as an increase in serum PSA that is ≥ 2 ng/mL above the nadir value observed following radiotherapy) or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Scott C Morgan, MD, MSc, Principal Investigator — The Ottawa Hospital Cancer Centre
Locations (1):
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No